CLINICAL TRIAL: NCT06288750
Title: Protective Effect of Indocyanine Green Fluorescence Imaging Technology on Parathyroid Glands During Total Thyroidectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Linglong Yingcheng Hospital (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: sdllycyyqx001
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Total Thyroidectomy; Parathyroid Function Low Adverse Event; Parathyroid Glands--Diseases; Indocyanine Green
MeSH Terms: conditions — Parathyroid Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indocyanine green group (Experimental): Identification of parathyroid glands (PGs) Near-infrared (NIR) fluorescence visualization of PGs, for only experimental group
  Interventions: Device: Indocyanine Green
- Traditional surgery group (Active Comparator): Conventional means of identification and assessment of PGs are mainly based on surgeon-dependent identification of their anatomical location and appearance (color, shape, etc.) by the naked eye.
  Interventions: Device: No indocyanine green

INTERVENTIONS:
Device: Indocyanine Green — ICG is a fluorescent dye which binds tightly to plasma proteins and becomes confined to the vascular system.
  Other Names: Near Infrared Fluorescence Imaging
  Arms: Indocyanine green group
Device: No indocyanine green — Conventional means of identification and assessment of PGs are mainly based on surgeon-dependent identification of their anatomical location and appearance (color, shape, etc.) by the naked eye.
  Arms: Traditional surgery group

SUMMARY:
Accurate identification and evaluation of the parathyroid glands (PGs) intraoperatively is critical to reduce the incidence of postoperative hypoparathyroidism after total thyroidectomy. Near-infrared fluorescence imaging (NIFI), including the autofluorescence (AF) and indocyanine green fluorescence (ICGF) imaging, is a promising technique to protect PGs. This study aimed to assess whether the combined use of AF and ICGF could reduce the incidence of postoperative hypoparathyroidism and improve the identification and evaluation of PGs during total thyroidectomy.

DETAILED DESCRIPTION:
Postoperative hypoparathyroidism or hypocalcemia is the most frequent complication after total thyroidectomy (TT) . The median incidence of transient and permanent postoperative hypoparathyroidism is 27% (19%-38%) and 1% (0-3%), respectively. Transient hypoparathyroidism can increase the length of hospital stay and the costs of hospitalization for patients. Permanent hypoparathyroidism leads to lifelong medication use, which may severely impair the quality of life of patients. Therefore, identifying the parathyroid glands (PGs) and preserving those with adequate blood perfusion intraoperatively has always been a crucial procedure during thyroidectomy.

Conventional means of identification and assessment of PGs are mainly based on surgeon-dependent identification of their anatomical location and appearance (color, shape, etc.) by the naked eye. However, this visual inspection is often influenced by the experience of the surgeon, intraoperative hemorrhage, ectopic PGs and so on, which makes it difficult to fully protect the PGs.

Currently, there has been an emergence of near-infrared fluorescence imaging (NIFI) that can be applied during thyroid or parathyroid surgery for the evaluation and identification of PGs. This technique mainly exploits the autofluorescence (AF) of PGs and indocyanine green fluorescence (ICGF ) imaging.PGs could exhibit stronger AF than the surrounding tissue under near-infrared light, which can be exploited to accurately identify PGs in real time. Subsequent studies have demonstrated that AF can not only detect PGs intraoperatively in real time and improve the intraoperative identification of PGs but also reduce the incidence of postoperative hypoparathyroidism. However, AF cannot assess the status of PG blood perfusion and consequently is not useful when determining whether PGs need to be autotransplanted.

Indocyanine green (ICG) fluorescence imaging may be a great solution to this problem. ICG is a safe fluorescent dye with fast metabolism and few adverse effects that can quickly combine with plasma proteins after intravenous injection and is widely used in angiography in multiple surgical disciplines. In recent years, several studies have shown that ICGF may be superior in evaluating blood perfusion and predicting the function of PGs in situ, subsequently guiding their autotransplantation. However, ICGF may not be very suitable for the identification of PGs before dissection, as the thyroid gland would also emit intense fluorescence after the injection of ICG, which may lead to difficulties in distinguishing them. Thus, AF and ICGF have their own advantages and disadvantages in the identification and evaluation of PGs, respectively. These two methods can be considered complementary.

In the present study, the investigators used AF in combination with ICGF imaging by one fluorescence imaging system during different steps of the surgical procedure. At the beginning of the operation, AF was used to identify the PGs before any dissection. Then, after the thyroid gland was removed, AF was used again to locate the PGs in situ. Finally, ICGF was applied to evaluate the blood perfusion of the PGs in situ and guide their autotransplantation. The aim of this randomized controlled trial was to assess whether this strategy could reduce the incidence of postoperative hypoparathyroidism and benefit the identification and evaluation of PGs during total thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged 18 years and above
* Scheduled for elective total or hemi thyroidectomy
* Normal liver and renal function
* No known hypersensitivity for iodine or ICG
* Able to understand the nature of the study procedures
* Willing to participate and give written informed consent

Exclusion Criteria:

* Age < 18 years
* Liver or renal insufficiency
* Known ICG, iodine, penicillin or sulfa hypersensitivity
* Pregnancy or breastfeeding
* Not able to understand the nature of the study procedure
* Not willing to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Identification of parathyroid glands (PGs) by NIR/ICG camera detected high-contrast | 1 year
  İntravenous injection of ICG dye, to identify PGs under NIR (High-contrast fluorescence seen or not)

SECONDARY OUTCOMES:
Central lymph node dissetion (CLND) | 1 year
  Number of positive lymph nodes (micrometastases)

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Qiu, MD, Principal Investigator — Shandong Linglong Yingcheng Hospital
Locations (1):
- Shandong Linglong Yingcheng Hospital, Yantai, Shandong, China

IPD SHARING:
Plan to Share IPD: No